CLINICAL TRIAL: NCT03174067
Title: Buprenorphine in the Emergency Department: Buprenorphine Versus Clonidine for Opioid Withdrawal
Brief Title: Buprenorphine in the Emergency Department
Acronym: BED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Health Centre Toronto (Other)
Responsible Party: Principal Investigator, Anita Srivastava, Staff Physician and Associate Professor, St. Joseph's Health Centre Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BED2013
Record Dates: First submitted 2017-05-24; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Opioid Withdrawal; Opioid-use Disorder
Keywords: buprenorphine; emergency department
MeSH Terms: conditions — Opioid-Related Disorders; Emergencies | interventions — Buprenorphine; Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Buprenorphine (Experimental): Patient receives buprenorphine in the emergency room based on a clinical trial protocol as well as a take home prescription for buprenorphine
  Interventions: Drug: Buprenorphine
- Clonidine (Active Comparator): Patient receives clonidine in the emergency room based on a clinical trial protocol and also receives a take home prescription for clonidine
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Buprenorphine — The participant receives buprenorphine
  Arms: Buprenorphine
Drug: Clonidine — The participant receives clonidine
  Arms: Clonidine

SUMMARY:
This is a pilot randomized control trial randomizing patients presenting in opioid withdrawal to the emergency department to receive either one of clonidine (usual standard of care) or buprenorphine for their opioid withdrawal. Primary treatment outcome is attendance at a rapid access addiction medicine clinic within a few days of emergency room presentation. Secondary treatment outcome is treatment status with respect to opioid agonist treatment at one month post emergency room visit.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting to the ED in opioid withdrawal or soon to be in withdrawal
2. Minimum age 16
3. English speaking
4. Active phone number
5. Ontario Health Insurance Program card

Exclusion Criteria:

1. Pregnant
2. Currently enrolled in a methadone or buprenorphine maintenance
3. Benzodiazepine addiction (or taking >50mg of valium equivalent/day)
4. Acute hepatitis or liver failure

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of participants attending the rapid access clinic | 2-5 days
  The number of participants who attend a rapid access clinic assessment after initial enrollment

SECONDARY OUTCOMES:
Number of participants who are on opioid agonist treatment | 30 days
  The number of participants who are maintained on some form of opioid agonist treatment at the one-month mark

CONTACTS AND LOCATIONS:
Overall Officials: Anita Srivastava, MD, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srivastava A, Kahan M, Njoroge I, Sommer LZ. Buprenorphine in the emergency department: Randomized clinical controlled trial of clonidine versus buprenorphine for the treatment of opioid withdrawal. Can Fam Physician. 2019 May;65(5):e214-e220. PMID 31088887